CLINICAL TRIAL: NCT06966167
Title: Comparison of Outcomes Between Femtosecond Laser-Assisted and Conventional Phacoemulsification in Fuchs Endothelial Corneal Dystrophy Patients With Cataracts
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jin Yang, Chief Physician, Eye & ENT Hospital of Fudan University
Other Study IDs: Fuchs FLACS vs CPS
Record Dates: First submitted 2025-05-03; First posted 2025-05-11 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Fuchs Endothelial Corneal Dystrophy; Cataract
Keywords: Fuchs Endothelial Corneal Dystrophy; Cataract; Femtosecond Laser-Assisted Cataract Surgery; Conventional Phacoemulsification Surgery
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- conventional phacoemulsification surgery (CPS)
- femtosecond laser-assisted cataract surgery (FLACS)

SUMMARY:
The goal of this observational study is to compare the mid- to long-term efficacy of femtosecond laser-assisted cataract surgery (FLACS) and conventional phacoemulsification surgery (CPS) in patients with moderate to severe Fuchs' endothelial corneal dystrophy (FECD) complicated by cataracts.

The main questions it aims to answer are:

Does FLACS lead to better preservation of corneal endothelial cells compared to CPS in patients with moderate to severe FECD? How do visual outcomes and corneal transparency compare between FLACS and CPS in this patient population?

Comparison Group:

Researchers will compare patients undergoing FLACS with those undergoing CPS to evaluate differences in endothelial cell loss, corneal thickness, visual acuity, and corneal transparency.

Participants:

Adults aged 40 years and older diagnosed with moderate to severe FECD (endothelial cell density <1500 cells/mm²).

Patients scheduled for cataract surgery at participating centers.

Participants will undergo:

Preoperative evaluations, including visual acuity tests, corneal endothelial cell density assessment (central and five peripheral zones), corneal thickness, and corneal densitometry.

Surgical intervention with either FLACS or CPS. Postoperative follow-ups at 1 day, 3 days, 1 week, 1 month, 3 months, 6 months, 1 year, and 2 years, including assessments of endothelial cell density, visual acuity, and corneal thickness.

This study aims to provide evidence-based recommendations for optimizing surgical strategies in high-risk patients with FECD and cataracts.

DETAILED DESCRIPTION:
Fuchs' endothelial corneal dystrophy (FECD) is a progressive, bilateral corneal disorder characterized by endothelial cell loss, Descemet's membrane thickening, and corneal edema, leading to visual impairment. Patients with moderate to severe FECD are particularly vulnerable to corneal decompensation following cataract surgery due to their compromised endothelial function. As cataract surgery is a common necessity in this patient population, selecting an appropriate surgical technique that minimizes endothelial cell damage is crucial to ensuring optimal postoperative outcomes.

This observational, prospective, multi-center controlled study aims to compare the mid- to long-term efficacy and safety of femtosecond laser-assisted cataract surgery (FLACS) versus conventional phacoemulsification surgery (CPS) in patients with moderate to severe FECD undergoing cataract extraction. The study seeks to determine which technique better preserves corneal endothelial integrity and maintains visual function, providing valuable insights into surgical decision-making for this high-risk patient population.

Study Objectives The primary objective of this study is to evaluate the differences in corneal endothelial cell density (ECD) loss and corneal thickness changes between FLACS and CPS in patients with moderate to severe FECD undergoing cataract surgery.

The secondary objectives include:

Assessing differences in postoperative visual acuity, including uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA).

Comparing corneal densitometry and transparency changes between the two surgical techniques.

Evaluating postoperative corneal edema and potential complications related to endothelial decompensation.

Study Design Type: Prospective, observational, multi-center, controlled study Study Sites: Three ophthalmology centers with similar surgical and imaging equipment Participants: 120 eyes from 120 patients (FLACS group: 80 eyes; CPS group: 40 eyes)

Grouping: Patients will be assigned to either FLACS or CPS based on clinical indications rather than randomization. Subgroup analyses will be conducted based on:

Age (>70 years vs. ≤70 years) Preoperative endothelial cell density (<1000 cells/mm² vs. ≥1000 cells/mm²) Cataract nuclear grading (>grade 3 vs. ≤grade 3) Eligibility Criteria

Inclusion Criteria:

Patients scheduled for cataract surgery Age ≥40 years Diagnosed with moderate to severe FECD (endothelial cell density <1500 cells/mm²)

Exclusion Criteria:

History of prior intraocular surgery Presence of ocular conditions other than FECD and cataracts (e.g., severe dry eye, corneal scarring, keratoconus, uveitis, uncontrolled glaucoma, vitreoretinal disease) Requirement for additional intraocular procedures during the study period (excluding Nd:YAG posterior capsulotomy)

Discontinuation Criteria:

Failure to complete scheduled follow-up visits Serious adverse events (e.g., vision-threatening endophthalmitis) Participant withdrawal from the study Interventions & Assessments

Preoperative Evaluation:

Comprehensive ophthalmic examination, including visual acuity testing (UDVA, CDVA), intraocular pressure (IOP), and refraction Biometric assessment using IOLMaster Corneal endothelial cell density measurement using specular microscopy and confocal microscopy (central, superior, inferior, nasal, and temporal zones) Corneal pachymetry and densitometry evaluation using Pentacam

Surgical Interventions:

FLACS Group: Patients will undergo femtosecond laser-assisted cataract surgery, which includes laser-assisted corneal incisions, capsulotomy, and lens fragmentation, followed by phacoemulsification.

CPS Group: Patients will undergo conventional phacoemulsification with manual capsulorhexis and lens nucleus fragmentation using ultrasound energy.

Postoperative Follow-Up Schedule:

Patients will be followed up at 1 day, 3 days, 1 week, 1 month, 3 months, 6 months, 1 year, and 2 years postoperatively. At each follow-up visit, the following assessments will be performed:

Visual acuity (UDVA, CDVA) Intraocular pressure measurement Corneal endothelial assessment using specular and confocal microscopy Corneal pachymetry and densitometry using Pentacam Outcome Measures

Primary Outcomes:

Change in central corneal endothelial cell density (ECD) from baseline to postoperative time points Change in corneal thickness from baseline to postoperative time points

Secondary Outcomes:

Change in corneal densitometry (central, superior, inferior, nasal, temporal zones) Postoperative visual acuity outcomes (UDVA, CDVA) Rate of corneal edema and decompensation Incidence of surgical complications (e.g., intraoperative endothelial damage, postoperative corneal haze) Statistical Analysis Continuous variables will be expressed as mean ± standard deviation (SD) and analyzed using t-tests or ANOVA.

Categorical variables will be analyzed using Chi-square tests. Non-normally distributed data will be evaluated using the Mann-Whitney U test. Longitudinal changes will be assessed using repeated-measures ANOVA or Friedman's test.

Pearson correlation analysis will be used to evaluate relationships between variables.

A p-value < 0.05 will be considered statistically significant.

Ethical Considerations This study will be conducted in compliance with the Declaration of Helsinki and national ethical guidelines. Informed consent will be obtained from all participants prior to enrollment. Patient confidentiality will be maintained through anonymized data collection and storage. The study protocol has been reviewed and approved by the institutional ethics committee.

Significance of the Study This study will provide critical evidence on the optimal surgical approach for cataract patients with FECD, guiding clinicians in making evidence-based surgical decisions to improve visual outcomes and reduce endothelial cell loss in this vulnerable population. It may also contribute to refining surgical techniques and identifying best practices for preserving corneal endothelial health during cataract surgery in patients with pre-existing endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cataract surgery
* Age ≥40 years
* Diagnosed with moderate to severe FECD (endothelial cell density <1500 cells/mm²)

Exclusion Criteria:

* History of prior intraocular surgery
* Presence of ocular conditions other than FECD and cataracts (e.g., severe dry eye, corneal scarring, keratoconus, uveitis, uncontrolled glaucoma, vitreoretinal disease)
* Requirement for additional intraocular procedures during the study period (excluding Nd:YAG posterior capsulotomy)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 40 years or older, diagnosed with moderate to severe Fuchs endothelial corneal dystrophy (endothelial cell density < 1500 cells/mm²), and presenting with visually significant cataract.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change in central corneal endothelial cell density (ECD) from baseline to postoperative time points | From enrollment to the end of treatment at 2years
Change in corneal thickness from baseline to postoperative time points | From enrollment to the end of treatment at 2years

SECONDARY OUTCOMES:
Change in corneal densitometry (central, superior, inferior, nasal, temporal zones) | From enrollment to the end of treatment at 2years
Postoperative visual acuity outcomes (UDVA, CDVA) | From enrollment to the end of treatment at 2years

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and ENT hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lupardi E, Moramarco A, Cassini F, Febbraro S, Savini G, Fontana L. Corneal densitometry measurements comparison between anterior segment OCT and scheimpflug imaging. Int Ophthalmol. 2024 Sep 25;44(1):392. doi: 10.1007/s10792-024-03309-0. PMID 39320570
- [Background] Aiello F, Gallo Afflitto G, Ceccarelli F, Cesareo M, Nucci C. Global Prevalence of Fuchs Endothelial Corneal Dystrophy (FECD) in Adult Population: A Systematic Review and Meta-Analysis. J Ophthalmol. 2022 Apr 14;2022:3091695. doi: 10.1155/2022/3091695. eCollection 2022. PMID 35462618
- [Background] Ali M, Cho K, Srikumaran D. Fuchs Dystrophy and Cataract: Diagnosis, Evaluation and Treatment. Ophthalmol Ther. 2023 Apr;12(2):691-704. doi: 10.1007/s40123-022-00637-1. Epub 2023 Jan 13. PMID 36637659
- [Background] Bourne WM, Nelson LR, Hodge DO. Central corneal endothelial cell changes over a ten-year period. Invest Ophthalmol Vis Sci. 1997 Mar;38(3):779-82. PMID 9071233